CLINICAL TRIAL: NCT05792124
Title: Comparison of the Effects of Retro Laminar Block (RLB) and Erector Spina Area Block (ESP) on Postoperative Recovery Quality and Pain in Lumbar Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, associate professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022/06
Record Dates: First submitted 2023-01-19; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pain
Keywords: Recovery Quality; postoperative pain; Erector spina plane block; Retrolaminar block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP BLOCK (Experimental)
  Interventions: Procedure: Erector spina area block
- RLB BLOCK (Active Comparator)
  Interventions: Procedure: Retrolaminar block

INTERVENTIONS:
Procedure: Erector spina area block — After anesthesia and surgical intervention, bilateral ESP passage will be performed with ultrasonography from the T10 level 3 cm lateral to the midline. After cleaning the area with povidone iodine before the block, T10 transverse output will be determined using a linear ultrasound probe. Local anesthetic will be applied to the erector spina with the use of the needle used for peripheral block procedures and transverse access. With the serum treatment from the local anesthesia application, the location of the needle will be correct with the hydrodissection method. After the location of the needle is confirmed, a mixture containing 20 ml of LA and serum will be applied and the same procedure will be repeated in the contralateral. 20 ml of total 40 ml LA is bupivacaine 0.5%, after 20 ml serum content.
  Arms: ESP BLOCK
Procedure: Retrolaminar block — The patient is in the prone position and the high-frequency linear ultrasound transducer is in parasagittal orientation, but the entry point is determined more medial than the ESP block. The needle entry point is 1-1.5 cm lateral to the targeted spinos process. The echogenic needle is advanced until it contacts the lamina in the craniocaudal plane and 0.5-1 for control. By giving cc 0.9 nacl solution, it is observed that the fluid is distributed between the erector spina muscle and the lamina. After the location of the needle is confirmed, a mixture of 20 ml of LA and saline will be applied and the same procedure will be repeated in the contralateral. 20 ml of total 40 ml LA will consist of bupivacaine 0.5% and 20 ml physiological saline.
  Arms: RLB BLOCK

SUMMARY:
The aim of this study is to compare the efficacy of erector spinae plane block (ESPB) and Retrolaminar Block on postoperative recovary quality and pain after lumbar spinal surgery

DETAILED DESCRIPTION:
The study was designed as a double-blind, prospective randomized controlled trial.

Blindness; The healthcare professionals who will monitor the patient's pain in the post-operative period will not know which of the ESP or RLB block is applied. Randomization of the patients was planned using computer aided. It was envisaged to include 40 participants each in the ESP block and RLB block groups. The current pain status of the patients in the ESP block and RLB block groups in the postoperative period was determined by NRS (Numerical rating scale) at rest and motion at certain hour intervals (30 .min,1.,6.,12.,24. hours) will be done, when the patients' NRS scores are 4 and above, an additional intravenous analgesic will be administered and the number of bolus doses with PCA in the first 24 hours will be recorded. The recovery quality of the patients who underwent both ESP block and RLB block at the postoperative 24th hour will be evaluated with a (QoR-40) scoring system. In addition, the hemodynamic values of the patients will be recorded in these intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar spinal surgery under elective conditions
* ASA I-III
* Between 18-75 ages

Exclusion Criteria:

* refuse during registration
* request to be dismissed from study
* failure to give informed consent
* emergency surgery
* bleeding diathesis
* Presence of contraindications to the LA agents used in this study chronic use of opioids psychiatric disorders the presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Qor-40 test (The recovery quality test) | 24th hour
  For this purpose, patients will be subjected to the Short Form-40- test, which is a short scale of postoperative recovery quality at first 24th hour.Minimum score is 40=bad ,maximum score is 200=good

SECONDARY OUTCOMES:
NRS (Numerical rating scale) | 30 minutes,1st hour,6th hour,12th hour and 24th hour
  It is a pain intensity determination system based on the system where the person tells a point between 0 =(no pain), 10= (unbearable pain) and to describe their pain.
Postoperative pain | 30 minutes,1st hour,6th hour,12th hour and 24th hour
  Postoperative opioid consumptions on the pca (patient controlled analgesia) device of the patients will be recorded in Postoperative 30.min,1.,6.,12.,24. Opioid consumptions on the pca device of the patients will be recorded in 30.min,1.,6.,12.,24. hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Faculty of Medicine, Aydin, Turkey (Türkiye)